CLINICAL TRIAL: NCT01832870
Title: Phase 1 Study of Sipuleucel-T and Ipilimumab in Combination for Advanced Prostate Cancer
Brief Title: Sipuleucel-T and Ipilimumab for Advanced Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prostate Oncology Specialists, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIPIPI 2013
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer; Castrate Resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Patients enrolled will receive the standard 3-dose treatment of sipuleucel-T, followed by treatment(s) of ipilimumab.
  Interventions: Drug: sipuleucel-T; Drug: ipilimumab

INTERVENTIONS:
Drug: sipuleucel-T
  Other Names: Provenge
Drug: ipilimumab
  Other Names: Yervoy

SUMMARY:
This is a clinical trial designed to quantify the immune response and determine the tolerability and side effects of sipuleucel-T when given in combination with ipilimumab for patients with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced prostate cancer who are eligible to receive sipuleucel-T in accordance with FDA approved labeling of sipuleucel-T
* Subjects must understand and sign an informed consent form

Exclusion Criteria:

* Subjects who are not eligible to receive sipuleucel-T

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Antigen-specific memory T cell response | After last sipuleucel-T and last ipilimumab, and follow-up period, an expected average of 15 months
  To quantify antigen-specific memory T cell response to sipuleucel-T and ipilimumab in combination.
Antigen-specific T cell proliferation to PA2024, PAP and PHA | After last sipuleucel-T and last ipilimumab, and follow-up period, an expected average of 15 months
  To quantify Antigen-specific T cell proliferation to PA2024, PAP and PHA when sipuleucel-T and ipilimumab are given in combination.
  * PA2024 is a recombinant protein
  * PAP: Prostatic acid phosphatase
  * PHA: Phytohaemagglutinin, an assay control
Antibody responses against PA2024 and PAP | After last sipuleucel-T and last ipilimumab, and the follow-up period, an expected average of 15 months
  To quantify antibody responses against PA2024 and PAP.
  * PA2024 is a recombinant protein
  * PAP: Prostatic acid phosphatase

SECONDARY OUTCOMES:
Prostate-Specific Antigen (PSA) doubling time | Duration of the study, an expected average of 18 months
  To measure changes in PSA doubling time following treatment with sipuleucel-T and ipilimumab
Time to PSA progression | Duration of the study, an expected average of 18 months
  To quantify time to PSA progression after treatment with sipuleucel-T and ipilimumab
Time to salvage therapy | Duration of the study, an expected average of 18 months
  To quantify time to salvage therapy after treatment with sipuleucel-T and ipilimumab
Percentage PSA decline | Duration of the study, an expected average of 18 months
  To measure percentage PSA decline following treatment with sipuleucel-T and ipilimumab

CONTACTS AND LOCATIONS:
Overall Officials: Mark Scholz, MD, Principal Investigator — Prostate Oncology Specialists, Inc.
Locations (1):
- Prostate Oncology Specialists, Inc., Marina del Rey, California, United States